CLINICAL TRIAL: NCT01498094
Title: A Prospective Open Randomized Clinical Trial Comparing High Flow Nasal Cannula Oxygen Therapy Against Standard Therapy for Children Hospitalized With Bronchiolitis
Brief Title: Study of High-flow Oxygen Therapy Against Standard Therapy in Bronchiolitis
Acronym: Hi-Flo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H11-03032
Record Dates: First submitted 2011-12-16; First posted 2011-12-23 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; High; Flow; Oxygen; Therapy; Nasal; Cannulae; Prongs
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Standard low-flow oxygen therapy.
  Interventions: Other: Standard low flow oxygen
- Intervention (Experimental): High Flow Nasal Cannula Oxygen Therapy
  Interventions: Procedure: High Flow Nasal Cannula Oxygen Therapy

INTERVENTIONS:
Procedure: High Flow Nasal Cannula Oxygen Therapy — Warm humidified oxygen will be delivered at 8 liters/minute via nasal cannulae, at a concentration that maintains saturations greater than 92%.
  Other Names: High flow oxygen therapy
  Arms: Intervention
Other: Standard low flow oxygen — Standard low flow oxygen will be given to patients to maintain saturations greater than 92%.
  Arms: Control

SUMMARY:
Bronchiolitis is a common illness of the respiratory tract caused by infection of the tiny airways within the lungs called bronchioles. At present the standard care of hospitalized children with bronchiolitis is oxygen via nasal prongs. In this study the investigators would like to compare standard ward management with a new method of delivering oxygen called high flow nasal cannula oxygen therapy (HFNOT). HFNOT involves breathing warmed, moistened oxygen through nasal cannulae at a flow rate of 8 liters/minute. Accumulated experience suggests that HFNOT eases the child's work of breathing and reduces need for ICU admission and invasive respiratory support.

DETAILED DESCRIPTION:
We propose a prospective open randomised controlled trial to compare high flow nasal cannula oxygen therapy (HFNOT) with standard oxygen therapy for infants hospitalised with bronchiolitis. This study will be the first of its kind, as currently there is no evidence in the published literature.

All children will be cared for by the same medical team on two wards. All aspects of care other than oxygen delivery will not be specified, and be at the discretion of the physicians. HFNOT will not be used as an escalation of care on the wards.

Randomisation will be performed by REDcap, in blocks of 6 patients. Patients will be identified in Emergency, informed consent obtained, and treatment started prior to transfer to the ward.

For patients randomised to HFNOT, the flow rate will be fixed at 8 liters/minute, and the inspired oxygen concentration titrated to maintain saturations above 92%.

Interim statistical analysis will be conducted to determine any positive or negative effect of HFNOT therapy. The first interval analysis will be performed after 50 subjects, the second after 100 subjects. If an effect is found, the study will be terminated following discussion with the hospital statistician and ethics board. Whichever treatment arm is found to be beneficial will be instituted as standard care for children with bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

* All children under 18 months of age with a clinical diagnosis of bronchiolitis requiring admission to hospital for observation and oxygen.

Exclusion Criteria:

* Infants admitted directly to ICU from Emergency.
* Prior positive pressure home ventilation.
* Tracheostomy.
* Nasogastric tubes in situ on admission.
* Upper airway abnormality.
* Congenital heart disease.

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2011-12; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Expected average length of stay 5 days
  Number of hours that the patient remains in hospital.

SECONDARY OUTCOMES:
Admission to Intensive Care Unit | During hospitalisation for bronchiolitis, expected average 5 days
  Yes or No
Work of breathing | During hospital stay, expected average 5 days
  Work of breathing, assessed by respiratory rate, at four timepoints on day one, and daily thereafter

CONTACTS AND LOCATIONS:
Overall Officials: David Wensley, MD, Principal Investigator — British Columbia Children's Hospital
Locations (1):
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada